CLINICAL TRIAL: NCT00238030
Title: Efficacy and Pharmacokinetics of Oral Thyroid Replacement Therapy in Organ Donors
Brief Title: Thyroxine Replacement in Organ Donors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr Michael D Sharpe, London Health Sciences Centre - University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-04-298
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Brain Death
Keywords: organ donation; thyroid replacement
MeSH Terms: conditions — Brain Death | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- po thyroxine (Active Comparator): placebo is iv
  Interventions: Drug: L-thryoxine; Drug: iv thryoxine
- iv thyroxine (Active Comparator): placebo is po
  Interventions: Drug: iv thryoxine

INTERVENTIONS:
Drug: L-thryoxine — 2 mcg/kg iv or 2 mcg/kg po at time of enrollment
  Other Names: L-thyroxine; Eltroxin
  Arms: po thyroxine
Drug: iv thryoxine — thyroxine 2 mcg/kg iv
  Other Names: L-thyroxine; Eltroxin

SUMMARY:
To compare oral versus intravenous administration of thyroid hormone: 1) for reversibility of hemodynamic instability in organ donors, and, 2) the pharmacokinetics of oral vs iv thyroid administration

DETAILED DESCRIPTION:
Disruption of the hypothalamic-pituitary axis following brain death may lead to hemodynamic instability, peripheral vasodilation, and diabetes insipidus in organ donors, requiring the use of high doses of inotropes. Inotropes may cause ischemic injury to organs and intramyocardial ATP stores, resulting in organs unsuitable for transplantation, as well as, a reduction in post-transplant organ function. Therefore, some clinicians advocate the use of triple hormonal therapy in potential organ donors.

Since intravenous T3(the intracellular active form of thyroxine) is unavailable, oral or intravenous T4 must be used, requiring the conversion of T4 to T3at the cellular level. This conversion is impeded by glucocorticoids which also are administered to organ donors for their immunomodulating effects. Since oral T3 is readily available, our first question is whether oral versus intravenous administration of T4 is comparable. If so, our next study is to determine the efficacy of oral T3 versus oral T4. Our hypothesis is oral T3 is superior to oral T4.

Our study therefore will determine whether or not the oral route is suitable for administration of thyroid replacement therapy. The study will compare the pharmacokinetics of oral versus intravenous T4 administration in organ donors, as well as, determine its ability to wean intropes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Brain death criteria established
2. Consent for organ donation received

Exclusion Criteria:

1. immediate (< 4 Hrs) organ retrieval anticipated

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-12; Primary Completion 2009-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Percentage of time patients require inotropic support prior to organ procurement. | every hour following administration

SECONDARY OUTCOMES:
pharmacokinetic profiles of oral vs iv T3,T4 | hourly from time of administration
number of organs donated | total number of organs donated at time of procurement
thyroid function derangements at time of brain death | thyroid function q 4hrs following declaration of brain death

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Sharpe, MD FRCPC, Principal Investigator — London Health Sciences Centre-UC+
Locations (1):
- London Health Sciences Centre-UC, London, Ontario, Canada

REFERENCES:
- [Background] Novitzky D, Cooper DK, Chaffin JS, Greer AE, DeBault LE, Zuhdi N. Improved cardiac allograft function following triiodothyronine therapy to both donor and recipient. Transplantation. 1990 Feb;49(2):311-6. doi: 10.1097/00007890-199002000-00017. PMID 2305461
- [Derived] Sharpe MD, van Rassel B, Haddara W. Oral and intravenous thyroxine (T4) achieve comparable serum levels for hormonal resuscitation protocol in organ donors: a randomized double-blinded study. Can J Anaesth. 2013 Oct;60(10):998-1002. doi: 10.1007/s12630-013-0004-x. Epub 2013 Jul 25. PMID 23884915